CLINICAL TRIAL: NCT07031466
Title: Treatment Outcome in Patients After eCPR
Status: Completed | Type: Observational
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Other Study IDs: FNO-KARIM-eCPR
Record Dates: First submitted 2025-06-12; First posted 2025-06-22 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Cardiac Arrest (CA)
Keywords: extracorporeal membrane oxygenation (ECMO); extracorporeal cardiopulmonary resuscitation (eCPR); Quality of Life; out-of-hospital cardiac arrest (OHCA); Post-Intensive Care Syndrome (PICS)
MeSH Terms: conditions — Heart Arrest; Out-of-Hospital Cardiac Arrest; postintensive care syndrome | interventions — Quality of Life

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective eCPR group: Retrospective analysis of eCPR patients
  Interventions: Other: Retrospective analysis of assigned treatment
- Prospective eCPR group: Prospective analysis of eCPR patients
  Interventions: Other: Quality of Life (SF-36); Other: Quality of Life (EQ-5D); Other: Hospital Anxiety and Depression (HADS)

INTERVENTIONS:
Other: Retrospective analysis of assigned treatment — Retrospective analysis of assigned treatment will be performed
  Groups: Retrospective eCPR group
Other: Quality of Life (SF-36) — The quality of life will be assessed using the SF-36 (Short-Form Health Subject Questionnaire).
  Groups: Prospective eCPR group
Other: Quality of Life (EQ-5D) — The quality of life will be assessed using the EQ-5D (European Quality of Life Questionnaire)
  Groups: Prospective eCPR group
Other: Hospital Anxiety and Depression (HADS) — Hospital Anxiety and Depression will be assessed using the HADS (Hospital Anxiety and Depression Scale)
  Groups: Prospective eCPR group

SUMMARY:
This study consists of two parts - retrospective and prospective. The aim of this study is to assess the quality of life in bio-psycho-social dimensions in patients after eCPR (extracorporeal cardiopulmonary resuscitation), in relation to their neurological outcome after the end of treatment and discharge from the Ostrava University Hospital (FNO). The study will focus on patients who underwent extracorporeal membrane oxygenation (ECMO) support after out-of-hospital cardiac arrest (OHCA) in the years 2022-2024.

DETAILED DESCRIPTION:
Retrospective study Quantitative evaluation using data analysis from documentation. Patients on ECMO after OHCA in the period 1. 1. 2022 - 31. 12. 2024 will be evaluated based on data from the documentation. Analysis of data from the documentation of selected patients will be performed, evaluating demographic data, comorbidities, duration of ECMO support, mortality, Cerebral Performance Category (CPC) score 30 days after CPR.

Prospective study Quantitative assessment using validated questionnaire tools Patients connected to ECMO after OHCA in the period 1. 1. 2022 - 31. 12. 2024, in whom a CPC score >3 was detected after the 30th day from cardiac arrest and who were discharged from the FNO. As part of patient dispensary, these patients are electively invited to the PICS outpatient clinic in the FNO Ostrava. Individual interviews (filling out questionnaires) will be performed after obtaining informed consent in the Post-Intensive Care Syndrome (PICS) outpatient clinic at the University Hospital Ostrava, or telephone interviews conducted by the attending physician.

ELIGIBILITY:
Inclusion Criteria:

* Patient who underwent eCPR after OHCA at University Hospital Ostrava
* Hospitalised in the period from 1. 1. 2022 to 31. 12. 2024
* Ability to undergo an interview personally or a family member able to provide information
* Signed informed consent

Exclusion Criteria:

* Language barrier
* Acute serious mental or somatic disease making the interview not feasible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent eCPR at the University Hospital Ostrava
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Quality of Life (SF-36) | 30 days
  Quality of Life in patients after eCPR will be assessed using the SF-36 questionnaire 30 days after eCPR
Quality of Life (EQ-5D) | 30 days
  Quality of Life in patients after eCPR will be assessed using the EQ-5D questionnaire 30 days after eCPR
Hospital Anxiety and Depression Scale (HADS) | 30 days
  Hospital Anxiety and Depression Scale (HADS) in patients after eCPR will be assessed using the EQ-5D questionnaire 30 days after eCPR

CONTACTS AND LOCATIONS:
Overall Officials: Michaela Lišková, Bc., Principal Investigator — University of Ostrava
Locations (2):
- Czechia (2):
  - University of Ostrava, Ostrava, Moravian-Silesian Region
  - University Hospital Ostrava, Ostrava, Moravian-Silesian Region

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers. The data may be provided upon request.